CLINICAL TRIAL: NCT00277953
Title: A Review of Tracheal Dimensions in the Pediatric Population Using MRI
Brief Title: MRI Review of Tracheal Dimensions
Status: Terminated | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 04-047
Record Dates: First submitted 2006-01-13; First posted 2006-01-18 (Estimated); Last update posted 2007-05-04 (Estimated); Status verified 2007-05

CONDITIONS: Congenital Disorders
Keywords: Pediatric; Cardiac; Tracheal Dimensions; MRI
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

SUMMARY:
To date, there have been no published reports of normal variations in tracheal dimensions for pediatric patients undergoing MRIs. While there are reports of normals in CT studies, the reported dimensions were for average areas and lengths over the entire length of the trachea and not for normal variation in the dimensions at various sites in the trachea. Moreover, CT measurements are likely not entirely applicable to MRI measurements. Since cardiac MRI has become the procedure of choice to document the presence of vascular rings as well as the significance of any ring that is found, there is a need for normal values to be generated. This would in turn permit physicians to determine in cases of documented vascular rings the severity of the tracheal stenosis/deformity if found.

DETAILED DESCRIPTION:
To date, there have been no published reports of normal variations in tracheal dimensions for pediatric patients undergoing MRIs. While there are reports of normals in CT studies, the reported dimensions were for average areas and lengths over the entire length of the trachea and not for normal variation in the dimensions at various sites in the trachea. Moreover, CT measurements are likely not entirely applicable to MRI measurements. Since cardiac MRI has become the procedure of choice to document the presence of vascular rings as well as the significance of any ring that is found, there is a need for normal values to be generated. This would in turn permit physicians to determine in cases of documented vascular rings the severity of the tracheal stenosis/deformity if found.

Hypothesis: Patients referred for cardiac MRIs to evaluate vascular rings will have significantly smaller tracheal dimensions (area, longest width, shortest width) based on a percentage of their maximal tracheal dimension in comparison with patients referred for cardiac MRIs for other indications.

I would propose to retrospectively review cardiac MRIs for tracheal dimensions in 25 consecutive patients referred for possible vascular rings and for 50 consecutive patients undergoing cardiac MRIs for other indications. As part of this study I would also propose to review the clinical findings that prompted the cardiac MRI to be ordered (i.e. respiratory symptoms, abnormal echocardiogram, abnormal CXR or barium swallow).

ELIGIBILITY:
Inclusion Criteria:

* 25 consecutive patients referred for possible vascular rings 50 consecutive patients undergoing cardiac MRIs for other indications adequate axial double-inversion recovery images of sufficient quality to permit accurate measurement of variations in tracheal dimension.

Exclusion Criteria:

* Those who do not meet inclusion criteria

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75

CONTACTS AND LOCATIONS:
Overall Officials: Denver Sallee III, MD, Principal Investigator — Children's Healthcare of Atlanta, Sibley Heart Center Cardiology
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States